CLINICAL TRIAL: NCT07206485
Title: EFFECT OF VIBROACOUSTIC THERAPY DEVICE WITH LASER MOTION GUIDANCE ON BALANCE SENSORY INTEGRATION IN PATIENTS WITH STROKE
Brief Title: VIBROACOUSTIC THERAPY in PATIENTS WITH STROKE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Assistant Professor of Neurology and Neurosurgery Faculty of Physical Therapy October 6 University, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/0
Record Dates: First submitted 2025-09-19; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group (I) (Experimental): will receive vibroacoustic therapy and a selected physical therapy program.
  Interventions: Device: vibro-acoustic therapy; Other: selected physical therapy exercises program
- Group (II) (Experimental): laser motion guidance therapy and a selected physical therapy program
  Interventions: Device: Motion Guidance Laser; Other: selected physical therapy exercises program
- Group (III) (Experimental): vibroacoustic therapy, laser motion guidance and a selected physical therapy program
  Interventions: Device: vibro-acoustic therapy; Device: Motion Guidance Laser; Other: selected physical therapy exercises program
- Group (IV) (Experimental): the selected physical therapy program
  Interventions: Other: selected physical therapy exercises program

INTERVENTIONS:
Device: vibro-acoustic therapy — Vibroacoustic therapy (VAT) is a type of sound therapy that involves passing low frequency sine wave vibrations into the body via a device with embedded speakers
  Arms: Group (I); Group (III)
Device: Motion Guidance Laser — Motion Guidance Laser is a tool used to improve the curative progression by leading to excessive participation of the subject, helping to facilitate motor skills, postural stability
  Arms: Group (II); Group (III)
Other: selected physical therapy exercises program — 1. Passive Prolonged Stretching and positioning
  2. Range of motion exercises for both upeer limb and lower limb
  3. Balance exercises static and dynamic

SUMMARY:
PURPOSE: to investigate the effect of vibroacoustic therapy device with laser motion guidance affect balance sensory integration in patients with stroke BACKGROUND: Following stroke, motor recovery can be dictated by the degree of sensory disruption, The application of vibroacoustic therapy device with laser motion guidance could improve balance and sensory integration functions.

DETAILED DESCRIPTION:
Forty-four patients post vascular stroke, from both sexes were participated in this study. The patients were randomly divided into four equal groups; Group (I) will receive vibroacoustic therapy and a selected physical therapy program. Group (II) will receive laser motion guidance therapy and a selected physical therapy program. Group (III) will receive vibroacoustic therapy, laser motion guidance and a selected physical therapy program. Group (IV) will receive the selected physical therapy program. The evaluation methods by Biodex balance system using Clinical Test of Sensory Integration and Balance (CTSIB), Time up and go test, and The Functional Independence Measure

ELIGIBILITY:
Inclusion Criteria:

* Forty-four patients post vascular stroke, according to a sample size calculation
* Both genders (males and females) will participate in the study.
* The age of patients will be from 45 to 60 years.
* The duration of the stroke will be at least 6 months.

Exclusion Criteria:

* Other brain injuries/ illnesses, cognitive impairment, serious sensory impairment (superficial, deep, or cortical sensation) or proprioceptive loss, vestibular disorders
* Severe apraxia, severe aphasia
* contractures that restrict patients movement

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Biodex balance system | four weeks
  Clinical Test of Sensory Integration and Balance (CTSIB) The Biodex Balance System provides objective, computer-based measurements for the Clinical Test of Sensory Integration and Balance (CTSIB), also known as the Sensory Organization Test (SOT), by quantifying postural sway under various sensory conditions.
Time up and go test (TUG) | four weeks
  The TUG is a general physical performance test used to assess mobility, balance, and locomotor performance in elderly people
Biodex balance system Overall Stability Index (OSI) | four weeks
  The Biodex Overall Stability Index (OSI) is a composite measure of postural stability provided by the Biodex Balance System (BBS). It quantifies how well a person can maintain balance by measuring the total deviation of the foot platform from level in both anterior-posterior (front-to-back) and medial-lateral (side-to-side) directions

SECONDARY OUTCOMES:
The Functional Independence Measure (FIM) scale | four weeks
  The Functional Independence Measure (FIM) is a standardized assessment tool used in rehabilitation to measure a patient's functional ability and level of disability across 18 items, scored on a 1-7 scale, to track progress and guide care plans The FIM assesses a total of 18 items across six categories-self-care, sphincter control, mobility, locomotion, communication, and social cognition-each focusing on essential daily activities.